CLINICAL TRIAL: NCT01200147
Title: Effectiveness of Rupture of Schatzki's Ring Using Biopsy Forceps Versus SIngle Dilation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer stopped producing rings
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Schatzki-2010
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Dysphagia; Schatzki Ring
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study withdrawn no details (No Intervention)
  Interventions: Other: study withdrawn no details

INTERVENTIONS:
Other: study withdrawn no details

SUMMARY:
Dysphagia is a common reason for referal to the investigators Gastoenterology service. As many as 14% of patients undergoing radiological studies for dysphagia are found to have schatzki rings. Current recommendations for treatment of patients with symptomatic Schatzki rings are based on ancedotal experience and uncontrolled studies. The only randomized study on comparison of techniques the investigators were able to locate was published in 2000 and included only 26 patients. This study demonstrated that the biopsy techinque was as effective as and better tolerated than the standard dilation technique. Considering that the cost and time required for dilatation is greater than the basic biopsy technique, significant cost savings could be achieved using the biopsy technique. As well, patient satisfaction is an important factor considering that Schatzki rings can recur and repeated endoscopy is often required. Therefore, a study that shows a technique to be as or better than the current standard in effectiveness, cost, time, and patient comfort could lead to shift in current practice.

DETAILED DESCRIPTION:
None available, study was withdrawn

ELIGIBILITY:
Inclusion Criteria:

* Presenting to endoscopy unit with symptoms of dysphagia or known history of schatzki ring

Exclusion Criteria:

* Prior esophageal or gastric surgery, severe esophagitis, coagulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark McMillan, MD FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- VG Hospital-Capital District Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
study withdrawn, no patients enrolled